CLINICAL TRIAL: NCT02439541
Title: Safety and Efficacy of Human Umbilical-Cord-derived Mesenchymal Stem Cell Transplantation in Ischemic Cardiomyopathy
Brief Title: Human Umbilical-Cord-Derived Mesenchymal Stem Cell Therapy in Ischemic Cardiomyopathy
Acronym: UCMSC-Heart
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Ivy Institute of Stem Cells Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307-IVY-SC-001
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Ischemic Heart Disease; Heart Failure; Angina
Keywords: cellular therapy; Chronic ischemic heart disease; phase 1/2 clinical study; human umbilical cord mesenchymal stem cell; ischemic heart disease; allogeneic stem cell transplantation
MeSH Terms: conditions — Heart Failure; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCMSC group (Experimental): Patients in this arm received umbilical cord MSCs by intracoronary injection
  Interventions: Biological: UCMSC group
- Control group (No Intervention): Patients in this arm did not receive any intervention.

INTERVENTIONS:
Biological: UCMSC group — Human umbilical cord MSCs are transplanted by intracoronary infusion(1×10^7)
  Arms: UCMSC group

SUMMARY:
Phase I-II Clinical Trial-Safety and efficacy of umbilical cord derived mesenchymal stem cells (UC-MSCs) in patients with chronic heart ischemia cohort and perspective study.

DETAILED DESCRIPTION:
Phase I-II Clinical Trial-Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with chronic heart ischemia cohort and prospective study.

Forty patients will be selected and divided into two groups according to patients' willingness to stem cell treatment. The patients who are willing to receive stem cell transplantation will receive UC-MSCs by coronary injection. The patients in control group will not receive any intervention.

Every patient will maintain their standard treatment of chronic heart ischemia, with maximum tolerated dosage without side effects.

The day of infusion will be considered day zero. From that moment, followup will be divided into 0-1,1-3, 3-6, and 6-12 months.

Clinical results will be analyzed after completion of 12 months of followup.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 y
* No option for PCI or CABG (Angiographies evaluated by an independent interventional cardiologist).
* Maximal tolerable angina and heart failure medication
* NYHA functional classification (I-III)
* Signed informed consent

Exclusion Criteria:

* Severe liver or renal dysfunction or hemorrhagic diseases not suitable for PCI.
* Severe cerebral ischemic stroke or cerebral hemorrhage within 6 month.
* History with malignant disease within 5 y of inclusion or suspected malignity
* Severe heart failure (NYHA functional classification IV)
* Diminished functional capacity for other reasons such as COPD, alcoholic cardiomyopathy, or viral myocarditis
* Clinical significant anemia, leukopenia, leukocytosis,or thrombocythemia
* Clinical significant abnormal prothrombin or partial thromboplastin time or anticoagulation treatment that cannot be paused during treatment
* Patients with reduced immune response or treated with immunosuppressive medication
* Combined with severe infectious diseases
* Pregnant or fertile women
* Socially and mentally disabilities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number and nature of adverse events | Within the first year after intracoronary infusion
  Evidence for new clinical/biological abnormalities.
Incidence of major adverse coronary events (MACE) | Within the first year after intracoronary infusion
  Major adverse coronary events (MACE) were defined as cardiac death, non-fatal myocardial infarction, or rehospitalization for acute coronary syndrome and for congestive heart failure.

SECONDARY OUTCOMES:
Exercise Time and Level | Post cell transplantation: 1, 3, 6, 12 months
  Exercise time and level as assessed via six minute walk test.
Quantify myocardium perfusion measured by SPECT | Post cell transplantation: 6, 12 months
  The efficacy of UC-MSC treatment was quantified by the differences between the two groups and from baseline to 6 and 12 months in perfusion images, as measured by SPECT.
Assessment of heart function by left ventricular ejection fraction | Post cell transplantation: 1, 3, 6，12 months
  Change in left ventricular ejection fraction was assessed with echocardiography after cell implantation.
Clinical Improvement in NYHA Classification | 1 year
  The NYHA scale ranges from 1 (best)"Mild- no limitation of physical activity due to heart failure" to 4 (worst) "Severe-Unable to carry out any physical activity without discomfort due to heart failure".

CONTACTS AND LOCATIONS:
Overall Officials: Bing Liu, M.D, Study Chair — 307-IVY Translational Medicine Center; Xiaozhong Zhang, M.D, Principal Investigator — Department of cardiology,Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of cardiology,Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China